CLINICAL TRIAL: NCT00861185
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Assess the Safety and Efficacy of Four Weeks of Oral Senicapoc Administration on Exercise-Induced Asthma
Brief Title: Study to Assess Safety and Efficacy of Oral Senicapoc Administration on Exercise-induced Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icagen (Industry)
Responsible Party: Seth V. Hetherington, M.D. Sr. VP Clinical and Regulatory Affairs, Icagen, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICA-17043-18
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Exercise Induced Asthma
Keywords: bronchospasm; exercise asthma; inflammation; KCa3.1
MeSH Terms: conditions — Asthma, Exercise-Induced; Bronchial Spasm; Inflammation | interventions — senicapoc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Senicapoc (Experimental)
  Interventions: Drug: senicapoc
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: senicapoc — Loading Dose: 80 mg twice daily x 3 days Maintenance Dose: 40 mg daily for remainder of the treatment period (total 4 weeks)
  Other Names: ICA-17043
  Arms: Senicapoc
Drug: Placebo — Placebo looks identical to active study medication and will be dosed according to the same dosing regimen
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether 4 weeks of dosing with senicapoc alleviates exercise induced asthma symptoms.

DETAILED DESCRIPTION:
Based on the unmet medical need for new agents in the treatment of asthma and the role of KCa3.1 in the function of several different cell types involved in the inflammatory response, and the effects seen in an animal model of allergic asthma, it is reasonable to explore the utility of senicapoc, a KCa3.1 blocker, as a novel treatment of asthma. This study will test the ability of senicapoc to alleviate bronchospasm induced by an exercise challenge in subjects with asthma. Exercise challenge studies have been conducted for many currently approved asthma medications. Exercise challenge studies provide a controlled environment and test conditions to investigate the potential usefulness of novel study drugs for the treatment of asthma. This study will be the first to test the ability of senicapoc to reduce airway bronchospasm after exercise challenge, which is one clinically important manifestation of asthma seen in patients. In summary, with a demonstrated safety profile across a wide range of doses in humans and efficacy in an animal model of allergic bronchospasm and hyper-responsiveness, the initiation of exploratory studies of senicapoc for treatment of asthma is justified.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent to participate in the study as HIPAA authorization;
* Clinically acceptable medical history, physical examination, 12 lead ECG, vital signs, and clinical laboratory tests
* History of physician-diagnosed asthma according to Global Initiative for Asthma, AND exercise-induced asthma/ bronchoconstriction;
* Current treatment for asthma with short-acting inhaled beta-2-agonist ONLY;
* Baseline FEV1 >65% of predicted at Screen Visit 1;
* A 20% or greater drop in FEV1 following exercise challenge on at least two separate occasions prior to enrollment;
* Non-smoker (refrained from any tobacco usage, or any products containing nicotine, for 6 months prior to Day 1);

Exclusion Criteria:

* Subject who has experienced any allergic reaction to a drug which, suggests an increased potential for a hypersensitivity to senicapoc (e.g., clotrimazole);
* Previous ingestion of senicapoc (ICA-17043)
* Pregnant or lactating female;
* Condition that might interfere with the absorption, distribution, metabolism, and/or excretion of drugs; subjects who have had any previous gastrointestinal surgery, except appendectomy or cholecystectomy (if performed more than 90 days prior to Screening Visit 1) or a history of clinically significant active cardiovascular, neurologic, endocrine, hepatic, or renal disorders;
* Infectious illness, e.g. acute bacterial, acute and chronic parasitic, fungal infection or viral infection within 6 weeks prior to Screening Visit 1 or between Screening Visit 1 and Day 1 (Randomization).
* Treatment for conditions other than asthma with systemic corticosteroids within 1 month prior to Visit 1.
* Asthma exacerbation having necessitated treatment with inhaled corticosteroids within 6 weeks prior to study Screening Visit 1.
* History of severe asthma as defined by use of oral/injectable corticosteroids within the last 3 months and/or more than two bursts in the last year.
* Undergoing desensitization therapy unless on a maintenance dose for at least 3 months prior to entry and will continue as such throughout study participation.
* History of chronic pulmonary diseases other than asthma.
* Considering or scheduled to undergo any surgical procedure during the duration of the study;
* Ingestion of any investigational medication within 30 days prior to Screening Visit 1;
* A positive plasma alcohol, or urine cotinine test at Screening Visit 1;
* Use of the following asthma medications for the stated period prior to Screening Visit 1 and throughout the study:

  * Oral or parenteral corticosteroids within 3 months prior to Screening Visit 1
  * Inhaled corticosteroids (ICS) (e.g., budesonide, fluticasone propionate) within 1 month prior to Screening Visit 1
  * long acting beta agonists; leukotriene receptor antagonists; or anti-cholinergic agents (e.g. tiotropium) within the 2 weeks prior to Screening Visit;
* Use of antihistamines within 3 days prior to Screening Visit 1;
* Has a >10 pack-year history of smoking;
* Hypertension at screen (BP > 150/90), if deemed by Investigator to be unfit to complete exercise challenge testing;
* Screen QTc > 450 msec or ECG not suitable for QT measurement (e.g., poorly defined termination of T-wave);
* After exercise challenge test, subject not recovering to at least 90% of baseline FEV1 following administration of short-acting beta-2-agonist.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The change from baseline in the maximal percentage decrease in forced expiratory volume in one second (FEV1) after exercise | Week 2 and Week 4

SECONDARY OUTCOMES:
- Area under the curve (AUC) for FEV1 after exercise challenge, - the length of time for recovery of FEV1 after exercise challenge, - changes in non-challenge pulmonary function tests, and an asthma control questionnaire. | Week 2 and Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon Stocker, Ph.D., Study Director — Icagen
Locations (9):
- United States (9):
  - Huntington Beach, California
  - Orange, California
  - Normal, Illinois
  - Metairie, Louisiana
  - St Louis, Missouri
  - Skillman, New Jersey
  - North Syracuse, New York
  - Canton, Ohio
  - Seattle, Washington